CLINICAL TRIAL: NCT06523673
Title: Stereotactic Body Radiotherapy (SBRT) for Oligo-Progression During First-Line Chemotherapy in Metastatic Non-Small Cell Lung Cancer (OPPRESS):A Randomized, Controlled, Open-label, Multi-Center Phase 3 Study
Brief Title: Stereotactic Body Radiotherapy for Oligo-Progression Metastatic Non-Small Cell Lung Cancer
Acronym: OPPRESS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPPRESS
Record Dates: First submitted 2024-06-28; First posted 2024-07-26 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Metastatic Non-Small Cell Lung Cancer; NSCLC Stage IV; OligoProgressive Metastatic Disease
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT arm (Experimental): SBRT is administered to the site of progression. During SBRT treatment, maintenance therapy was with ICI or bevacizumab or combined single-agent chemotherapy. After the occurrence of progression that is no longer suitable for SBRT treatment, switch to second-line systemic therapy (same as SOC).
  Interventions: Radiation: Stereotactic Body Radiotherapy; Drug: second-line systemic therapy
- SOC arm (Active Comparator): Second-line systemic therapy is based on docetaxel or albumin-paclitaxel. The combination of immunotherapy or anti-vascular drugs is evaluated by the study physician. The specific drug regimen is determined in conjunction with the patient's wishes. Palliative radiotherapy is acceptable.
  Interventions: Drug: second-line systemic therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy — The dose of radiation therapy is determined by the radiologist based on the clinical parameters of the lesion, including tumor size and location. In most cases, radiotherapy fractionation regimens range from 27-30 Gy/3 Fractions or 30-50 Gy/5 Fractions, and appropriate radiotherapy doses covering 27-70 Gy/3-10 Fractions can also be selected by the radiologist based on radiation limitations of neighboring endangered organs.
  Other Names: SBRT; Stereotactic Ablative Radiotherapy (SABR)
  Arms: SBRT arm
Drug: second-line systemic therapy — a second-line docetaxel/albumin-bound paclitaxel-based systemic therapy regimen
  Other Names: docetaxel-based chemotherapy; albumin-bound paclitaxel-based chemotherapy; immunotherapy

SUMMARY:
The goal of this clinical trial is to learn if Stereotactic Body Radiotherapy (SBRT) can treat the oligo-progressive metastatic non-small cell lung cancer (NSCLC) after first-line chemotherapy. The main questions it aims to answer are:

Does SBRT improve progression-free survival in oligo-progressive metastatic non-small cell lung cancer after first-line chemotherapy? Does SBRT improve overall survival and quality of life in oligo-progressive metastatic non-small cell lung cancer after first-line chemotherapy?

Researchers will compare SBRT in combination with standard of care (SOC) and SOC only to see if SBRT works to treat oligo-progressive metastatic non-small cell lung cancer after first-line chemotherapy.

Participants will:

Take SBRT in combination with SOC or SOC only. Visit the clinic for checkups and tests as required by the study. Keep a diary of their symptoms and complete the quality of life assessment questionnaire.

DETAILED DESCRIPTION:
This study is a prospective, randomized, controlled, open-label, multi-center phase Ⅲ study of patients with stage IV NSCLC who developed oligo-progression after prior first-line chemotherapy with clinical benefit lasting for ≥3 months, aiming to evaluate the efficacy and safety of applying SBRT to treat oligo-progressive NSCLC.

NSCLC patients with oligo-progression (≤5 extracranial progression sites) after ≥3 months of clinical benefit by first-line systemic therapy and who are suitable for SBRT will be screened to meet the enrollment criteria after signing the informed consent and will be randomized to the SBRT/standard of care (SOC) groups according to the stratification ratio of 1:1.

SBRT group: SBRT was performed on the progressive sites. During SBRT treatment, maintenance therapy was with ICI or bevacizumab or combined single-agent chemotherapy. Evaluation was performed after completion of SBRT treatment. After the occurrence of progression that is no longer suitable for SBRT treatment, switch to second-line systemic therapy (same as SOC).

SOC group: Second-line systemic therapy is based on docetaxel or albumin-paclitaxel. The combination of immunotherapy or anti-vascular drugs is evaluated by the study physician. The specific drug regimen is determined in conjunction with the patient's wishes. Palliative radiotherapy is acceptable.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years. Gender is not limited.
* Histologically and/or cytologically confirmed stage IV metastatic NSCLC.
* Eastern Cooperative Oncology Group (ECOG) score of 0-2.
* Patients who had prior first-line chemotherapy with clinical benefit lasting for ≥3 months.
* Driver gene-negative NSCLC patients with oligo-progression during first-line chemotherapy combined with Immune Checkpoint Inhibitors (ICI). Driver gene-positive NSCLC patients, such as epidermal growth factor receptor (EGFR) mutation or anaplastic lymphoma kinase (ALK) fusion positivity, are allowed to enroll if oligo-progression occurred during treatment with first-line chemotherapy combined with bevacizumab ± ICI after failure of Tyrosine Kinase Inhibitor (TKI) therapy.
* Progressive sites were assessed as ≤5 according to RECIST v1.1 criteria combined with positron emission tomography / computertomography (PET/CT), and all were located extracranially. Progressive lymph node lesions are counted by region, with each lymph node region amenable to concurrent SBRT (which may contain multiple progressive lymph nodes) counted as 1 progressive site.
* All progressive sites should be visible on radiologic imaging and assessed as suitable for SBRT treatment by a radiotherapist.
* Intracranial progressive lesions and symptomatic lesions can be treated with palliative radiotherapy and local therapy prior to enrollment and are not counted within the oligo-progressive sites.
* Expected survival time greater than 3 months.
* Comprehensive examination completed within 28 days prior to enrollment in the study and a complete blood count/differential, collected within 15 days, showing that the patient has normal internal organ function and normal bone marrow function.
* Negative serum or urine pregnancy test in females of childbearing age within 14 days prior to study enrollment.
* Patients are willing to provide written informed consent and must be willing to adhere to the prescribed follow-up schedule.

Exclusion Criteria:

* Currently participating in an interventional clinical study treatment that may affect this study, or have been treated with another investigational drug or investigational device that may affect this study within 4 weeks prior to first treatment.
* Pregnant or lactating women.
* Progression sites deemed unsuitable for SBRT treatment as assessed by radiotherapy specialists.
* Presence of untreated intracranial metastases or symptomatic progressive sites.
* History of malignancy other than NSCLC or untreated primary malignancy within the past 3 years.
* Serious active comorbidities that would interfere with treatment in this study.
* History or evidence of disease that could interfere with the results of the trial, prevent the subject from participating in the study throughout, abnormal values of treatment or laboratory tests, or other conditions that, in the opinion of the investigator, make enrollment inappropriate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | Time from date of randomization until the date of first documented progression or date of death from any cause after the second-line treatment, whichever came first, assessed up to 18 months.
  Progression-free survival, PFS: Time from date of randomization until the date of first documented progression or date of death from any cause after the second-line treatment, whichever came first.

SECONDARY OUTCOMES:
Overall Survival (OS) | Time from date of randomization to death (from any cause), assessed up to 36 months.
  Overall Survival，OS: Time from date of randomization to death (from any cause).
Quality of Life (QoL) | From enrollment to the end of survival follow-up at 36 months.
  Patient quality of life will be assessed using the patient-reported European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) - Core 30 (EORTC QLQ-C-30) scale. Patient-reported EORTC-QLQ-C30 scale results will be scaled and scored according to the procedures recommended by the EORTC Quality of Life Panel, and scale scores for each visit period of the trial will be analyzed, as well as change values relative to baseline.
Safety of SBRT | From enrollment to the end of treatment at 4 weeks
  the safety of SBRT

CONTACTS AND LOCATIONS:
Overall Officials: Fuming Qiu, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No